CLINICAL TRIAL: NCT00296790
Title: Ambien CR vs. Placebo For Treatment Of Insomnia Associated With Anxiety When Used Concomitantly With Escitalopram (Lexapro)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PM_L_0167
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-10

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

INTERVENTIONS:
Drug: zolpidem tartrate

SUMMARY:
A comparison of Zolpidem Tartrate Extended-Release (Ambien CR)vs. Placebo in the Treatment of Insomnia Associated with Generalized Anxiety Disorder (GAD) when Used Concomitantly with Escitalopram (Lexapro - antidepressant).

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male or female between the ages of 21and 64 years, inclusive;
2. Women must use a medically acceptable form of contraception during the entire study period, or: be surgically sterilized, post-menopausal, agree to use double-barrier contraception throughout the study period, or must have a negative urine pregnancy test prior to randomization;
3. Must meet the diagnostic requirements of Generalized Anxiety Disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders;
4. Score at least 18 on the Hamilton Rating Scale for Anxiety (HAM-A)
5. Must be either newly diagnosed or show symptoms of relapse during a period of no drug therapy for anxiety.
6. Subject must experience sleep disturbances at least three nights per week, for at least one month prior to study entry, based on historical data.
7. Subject must be stabilized on all long-term medication therapy for at least one month prior to study entry.

EXCLUSION

1. History of Post-Traumatic Stress Disorder;
2. Concomitant Major Depressive Disorder or Bipolar Disorder;
3. Any abnormal pre-study laboratory values that require clinical intervention
4. Shift work or requirement for a regular change in sleep schedule by at least six hours within the previous month.
5. Pregnant or breastfeeding
6. History of drug addiction, alcoholism, or drug abuse
7. Currently using a benzodiazepine or SSRI or more than 2 days of use within the 28 days preceding randomization.
8. A positive urine drug screen for compounds that would interfere with the assessment of a hypnotic.
9. Use of prescription and non-prescription sedative drugs;
10. Prior failure to respond to escitalopram therapy for anxiety
11. The presence of any untreated or uncompensated clinically significant renal, endocrine, gastrointestinal, hepatic, respiratory, cardiovascular, other neurologic, hematologic, oncologic, immunologic, cerebrovascular disease or malignancy.
12. History of sleep apnea
13. History of myasthenia gravis
14. Known hypersensitivity and/or allergy to or previous adverse experience with zolpidem or escitalopram or any of their excipients
15. Subject is currently participating in another clinical trial (or within 28 days of screening).

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 372
Dates: Start 2006-02; Study Completion 2007-02

PRIMARY OUTCOMES:
Evaluate safety and hypnotic efficacy of zolpidem tartrate extended release vs. placebo in treatment of insomnia associated with Generalized Anxiety Disorder when used concomitantly with escitalopram

SECONDARY OUTCOMES:
To show that treating insomnia from beginning of SSRI (Selective Serotonin Reuptake Inhibitor) treatment for anxiety results in improvement in quality of life and possibly greater response to anti-anxiety therapy

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States